CLINICAL TRIAL: NCT07163195
Title: Smart Bandage With App-Based Telemonitoring vs Standard Care for Venous Leg Ulcer: Randomized Trial
Brief Title: Smart Bandage With Telemonitoring vs Standard Care for Venous Leg Ulcer: Randomized Trial
Acronym: SMART-VLU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asmat Burhan (Other)
Responsible Party: Sponsor-Investigator, Asmat Burhan, Lecturer/Researcher, Faculty of Health Sciences, Universitas Harapan Bangsa, Universitas Harapan Bangsa
Organization: Universitas Harapan Bangsa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VLU-RCT-2025; B.LPPM.UHB/486/05/2025 (Other: Universitas Harapan Bangsa)
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Venous Leg Ulcer (VLU); Chronic Wound
Keywords: Venous Leg Ulcer; Chronic Wound; Smart Bandage; Telemonitoring; Digital Health; Mobile Application; Wound Care; Wound Healing; Randomized Controlled Trial; Indonesia
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to either the intervention group (smart bandage plus standard wound care) or the control group (standard wound care alone). Both groups will be followed for 12 weeks in parallel. Randomization will use computer-generated block randomization with allocation concealment. Outcome assessors and data analysts will be blinded to group assignments.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors who evaluate digital wound images and statistical analysts will be blinded to treatment allocation. Participants, care providers, and investigators will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Bandage + Standard Wound Care (Experimental): Participants in this arm will receive a smart bandage with integrated sensors (pH, temperature, and moisture) connected to a mobile telemonitoring platform. Wound data will be transmitted securely to wound care nurses for review. In addition, patients will receive standard wound care including compression therapy, conventional dressings, sharp debridement when indicated, and patient education.
  Interventions: Device: Smart Bandage with Telemonitoring
- Conventional Bandage + Standard Wound Care (Active Comparator): Participants will receive standard wound care (compression therapy, debridement when indicated, and patient education) plus a conventional bandage without digital monitoring features. This represents usual care according to international guidelines
  Interventions: Device: Conventional Bandage

INTERVENTIONS:
Device: Smart Bandage with Telemonitoring — A smart wound bandage with integrated sensors (pH, temperature, moisture) connected to a mobile telemonitoring platform. Wound data are transmitted securely to a mobile application monitored by wound care nurses. The device is applied in addition to standard wound care (compression therapy, conventional dressing, debridement when indicated, and patient education).
  Other Names: Smart wound bandage, Digital wound monitoring bandage
  Arms: Smart Bandage + Standard Wound Care
Device: Conventional Bandage — A conventional wound bandage without digital monitoring features. It is applied in addition to standard wound care (compression therapy, conventional dressing, debridement when indicated, and patient education). This represents usual care according to international guidelines.
  Other Names: Standard wound dressing, Non-digital bandage
  Arms: Conventional Bandage + Standard Wound Care

SUMMARY:
Venous leg ulcers (VLUs) are chronic wounds that are often slow to heal and can greatly affect patients' daily lives. This study will evaluate a new "smart bandage" that can monitor wound conditions such as pH, temperature, and moisture, and transmit this information to a mobile app for nurses to review. Care can then be adjusted in real time.

The purpose of this randomized controlled trial is to compare smart bandage plus standard wound care with standard wound care alone. We will assess whether the smart bandage improves healing rates within 12 weeks, shortens time to healing, reduces infection, and improves quality of life in patients with VLUs. About 110 adult participants with VLUs will be enrolled at Clinic Podiatry Care, Purwokerto, Indonesia.

DETAILED DESCRIPTION:
Venous leg ulcers (VLUs) are chronic wounds with significant clinical and economic burden. Healing is often delayed due to persistent inflammation, tissue hypoxia, and susceptibility to infection. Smart bandage technologies offer a novel approach by integrating sensors that can continuously monitor wound conditions (pH, temperature, moisture) and transmit data via a mobile application for real-time telemonitoring. This enables wound care providers to adjust treatment promptly and may improve patient engagement and outcomes.

This randomized controlled trial will compare smart bandage plus standard wound care with standard wound care alone in adult patients with VLUs. The intervention group will receive a smart bandage with pH, temperature, and moisture sensors connected to a secure mobile app monitored by wound care nurses. The control group will receive standard care including compression therapy, conventional dressings, debridement as indicated, and patient education.

The primary outcome is the proportion of ulcers achieving complete healing within 12 weeks, defined as full epithelialization without drainage. Secondary outcomes include time to healing, percentage wound area reduction (measured by digital planimetry), incidence of clinical infection, and health-related quality of life (Wound-QoL questionnaire). A total of 110 participants will be recruited at Clinic Podiatry Care, Purwokerto, Indonesia.

Randomization will be performed in a 1:1 ratio using computer-generated block randomization. Outcome assessors and data analysts will be blinded. Analyses will follow the intention-to-treat principle, with χ² tests for primary outcomes and generalized estimating equations for repeated measures.

The study is designed to provide robust clinical evidence on the effectiveness of smart bandage technology combined with telemonitoring in VLU care, with the potential to inform integration of digital wound care into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years
* Clinically diagnosed venous leg ulcer persisting for more than 3 weeks
* Able to provide written informed consent

Exclusion Criteria:

* Age >65 years (elderly patients excluded)
* Acute or emergency wounds
* Mixed etiology ulcers with significant arterial involvement
* Severe comorbid illness such as end-stage renal failure or active malignancy
* Cognitive impairment preventing informed consent
* Allergy to dressing materials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of ulcers achieving complete healing | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Complete healing is defined as full epithelialization of the ulcer without drainage, confirmed at two consecutive visits by wound care nurses using standardized clinical assessment.

SECONDARY OUTCOMES:
Percentage reduction in wound area | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Change in ulcer size from baseline, measured using standardized digital photography and analyzed with ImageJ planimetry.
Health-related quality of life | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Wound Quality of Life questionnaire (Wound-QoL-17). Report global score and three subscales: Body/Physical, Psyche/Psychological, Everyday life. Scores are calculated as the mean item on a scale of 0-4; range 0-4, and higher scores = poorer quality of life (greater impairment). Reported as change from baseline at each time point.
  Unit of Measure: points (0-4)
Incidence of clinical infection | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Presence of infection determined by clinical signs and classified according to the Society for Vascular Surgery WIfI system.

CONTACTS AND LOCATIONS:
Overall Officials: Septian Mixrova Sebayang, MSN, Principal Investigator — Universitas Harapan Bangsa - Clinic Podiatry Care, Purwokerto
Locations (1):
- Podiatry Clinic, Banyumas, Indonesia, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) for primary and secondary outcomes, including baseline demographics, ulcer characteristics, intervention assignment, and outcome data.
  Time Frame:
  Available starting 6 months after publication of the main results, for up to 3 years.
  Access Criteria:
  Available to qualified researchers with sound proposals consistent with the study objectives.
  Access Method:
  By request to the Principal Investigator via email; access requires a data sharing agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: De-identified IPD and supporting information (study protocol, SAP, and analytic code) will be available beginning 6 months after publication of the main trial results and will remain available for 3 years thereafter.
Access Criteria: De-identified individual participant data (IPD) and supporting information (study protocol, SAP, and analytic code) will be made available to qualified researchers with methodologically sound proposals. Data will be provided for use in research consistent with the original trial objectives. Requests should be directed to the Principal Investigator via email. Access will be granted after review of the proposal and signing of a data sharing agreement.

REFERENCES:
- See also: Official study information page hosted by Klinik Podiatry Care, Purwokerto — https://u.podiatricare.my.id
- Available data/document: Individual Participant Data Set: Protocol_V1_2025 — https://u.podiatricare.my.id/ — The de-identified IPD underlying primary and secondary outcomes, along with the study protocol and SAP, will be available upon reasonable request to the Principal Investigator via email. Access requires a data sharing agreement.
- Available data/document: Statistical Analysis Plan: SAP_V1_2025 — https://u.podiatricare.my.id/ — The statistical analysis plan (SAP) describes predefined methods for analyzing the primary and secondary outcomes, including sample size justification, handling of missing data, and statistical tests. Available upon request to the PI
- Available data/document: Analytic Code: Code_V1_2025 — https://u.podiatricare.my.id/ — Analytic code used for data processing and statistical analyses, including scripts for wound area measurement (ImageJ) and outcome analyses (SPSS/R). The code will be available by request to the PI and requires a data sharing agreement